CLINICAL TRIAL: NCT01170819
Title: Double Balloon Catheter Versus Vaginal PGE2 for Pre-induction Cervical Ripening: a Randomized Study.
Brief Title: Double Balloon Catheter Versus Dinoprostone Vaginal Insert for Cervical Ripening.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonella Cromi, PhD, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1229
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Cervical Ripening; Labor Induction
Keywords: Cervical ripening; Induction of labor; Prostaglandins; Mechanical methods; Balloon catheter
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dinoprostone Vaginal Insert (Active Comparator)
  Interventions: Drug: Dinoprostone 10 mg controlled-release vaginal insert
- Double Balloon Catheter (Experimental)
  Interventions: Device: Double balloon catheter

INTERVENTIONS:
Device: Double balloon catheter — The balloons either side of the cervix are inflated with 50 ml of water. The catheter is removed after 12 hours if spontaneous expulsion has not occurred.
  Other Names: COOK CERVICAL BALLOON, COOK UROLOGICAL INC. US
  Arms: Double Balloon Catheter
Drug: Dinoprostone 10 mg controlled-release vaginal insert — Vaginal insert is placed in the posterior vaginal fornix for a maximum period of 24 hours.
  Other Names: PROPESS®, Ferring Pharmaceuticals
  Arms: Dinoprostone Vaginal Insert

SUMMARY:
To compare the efficacy of transcervical double balloon catheters versus controlled release dinoprostone vaginal inserts for pre-induction cervical ripening in term women with unfavourable cervices.

ELIGIBILITY:
Inclusion Criteria:

* singleton gestation
* gestational age greater than 34 weeks
* cephalic presentation
* intact membranes
* Bishop score of ≤4
* reactive fetal heart rate (FHR) pattern on admission

Exclusion Criteria:

* any condition precluding vaginal delivery
* any contraindication to receiving prostaglandins, including history of asthma, glaucoma, or cardiac or cardiovascular disease
* previous cesarean section or other uterine incision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Vaginal delivery within 24 hours | 24 hours from start of cervical ripening

SECONDARY OUTCOMES:
Cesarean section rate | 48 hours from start of ripening
Onset of active labor | 36 hours from start of ripening
  Active labor is defined as at least 4 uterine contractions in a 30 minutes interval with a totally effaced cervix and a cervical dilatation ≥3 cm
Uterine hyperstimulation | 12 hours (double ballon catheter arm) and 24 hours (dinoprostone vaginal insert arm) from start of ripening

CONTACTS AND LOCATIONS:
Locations (1):
- Del Ponte Hospital, Varese, Italy

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264